CLINICAL TRIAL: NCT04746508
Title: The Influence of Bilateral and Unilateral Flat Foot on Coronal Spinopelvic Alignment in Asymptomatic Young Healthy Males
Brief Title: Flat Foot and Coronal Spinopelvic Alignment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pınar Kısacık, PhD, Principle Investigator, Hacettepe University
Other Study IDs: 72300690-799-E17195
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Flat Foot [Pes Planus] (Acquired), Left Foot; Flat Foot [Pes Planus] (Acquired), Right Foot; Flat Foot Acquired Bilateral (Pes Planus); Pelvic Obliquity; Spinal Curvatures
Keywords: Flat foot; pelvic obliquity; spinal asymmetry; Cobb angle; calcaneal pitch angle
MeSH Terms: conditions — Flatfoot; Spinal Curvatures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unilateral Flat Foot (UniFF): Participants with flat foot unilaterally (Only one foot's Calcaneal pitch angle ≤ 20 degree)
- Bilateral Flat Foot (BiFF): Participants with flat foot bilaterally (Both feet's Calcaneal pitch angle ≤ 20 degree)

SUMMARY:
This study aimed to present the influence of unilateral and bilateral flat foot on coronal spinopelvic alignment in asymptomatic young healthy males. It will be carried out by examining the medical reports of individuals who apply to the National Health Board to work in positions requiring physical fitness between January 2018 and January 2019. Plain radiographies of the feet, pelvis, and spine will be analyzed. Calcaneal pitch angle (CPA) for flat foot, pelvic obliquity (PO), and Cobb angle (CA) for spinal asymmetry will be measured. After all analyzes were completed, participants will be divided into 2 groups as unilateral (UniFF) or bilateral (BiFF) flat foot, depending on the CPA measurements and will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ranging between 18.5-24.9 kg/m2 (accepted as normal weight by World Health Organisation (WHO))
* Age ranging between 18-25 years
* Male gender

Exclusion Criteria:

* Being older than 25 years
* BMI out of normal weight according to WHO
* Being female
* History of spinal trauma/ surgery
* Having/had spinal disorders like spondylolisthesis, spondylodiscitis, etc.
* Having/had chronic inflammatory arthritis especially spodiloarthrosis (i.e., ankylosing spondylitis, psoriatic arthritis, etc.)
* Having/had a vertebral fracture
* Having/had aseptic necrosis of the vertebra
* Radiographs with inappropriate image qualities.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy individuals who applied to the National Health Boards to work in positions requiring physical fitness between January 2018 and January 2019.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Calcaneal pitch angle (CPA) | Baseline
  Calcaneal pitch angle (CPA) is defined as an angle between a line drawn from the inferior of the calcaneocuboid joint to the inferior border of the calcaneus and a second line drawn from the inferior aspect of the sesamoid bones to the inferior border (13). CPA for both (right and left) foot was evaluated from all plain radiographs in this study and the angles equal to or less than 20 degrees were accepted as a flat foot.
Pelvic obliquity (PO) | Baseline
  Pelvic obliquity (PO) was measured by horizontal pelvic obliquity according to Osebold et al. from a posteroanterior radiograph. The angle between the line drawn between the most proximal points on the iliac crest and the line drawn parallel to the lower end of the radiograph was recorded.
The Cobb angle (CA | Baseline
  The Cobb angle (CA) is a gold standard measurement for identifying the magnitude of spinal curves (14). Spinal curvature was measured from the standing full-length posteroanterior radiograph. The angle of the curve is measured as an angle between the perpendiculars of the lines parallel to the upper border of the upper vertebral body and parallel to the lower border of the lowest vertebral body of the curve (16). Straight or symmetrical spines in the coronal plane were accepted as a normal spine, and curves<10 degrees accepted as spinal asymmetry, and the curves ≥ 10 degrees accepted as scoliosis (15). Spinal curve patterns in coronal planes were classified according to the Scoliosis Research Society classification. The curve was classified as single in terms of one curve exists in the thoracal or lumbal spine; as double in terms of one curve exist the through thoracal and lumbal spine; and as triple that exists through upper thoracal, middle thoracal and lumbal spine (17).

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kısacık, PhD, Principal Investigator — Hacettepe University Faculty of Physical Therapy and REhabilitation
Locations (1):
- Pınar Kısacık, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No